CLINICAL TRIAL: NCT00507234
Title: A 6-Week Trial to Compare the Efficacy and Safety of Concomitant Treatment With Formoterol Fumarate Inhalation Solution 20 Mcg Twice Daily and Tiotropium 18 Mcg Once Daily to Tiotropium 18 Mcg Once Daily Alone in the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Study in Subjects Greater Than 40 Years of Age With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201-080
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: formoterol fumarate inhalation solution

SUMMARY:
This is a multicenter, Phase IIIb, randomized, double-blind, active-controlled, parallel-group, comparative study.

The objectives of this study are:

1. To compare the efficacy of tiotropium 18 mcg once daily plus Formoterol Fumarate Inhalation Solution (FFIS) 20 mcg twice daily to tiotropium 18 mcg once daily.
2. To obtain safety data on the use of tiotropium 18 mcg once daily plus FFIS 20 mcg twice daily compared to tiotropium 18 mcg once daily.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of COPD
* Current or prior history of cigarette smoking

Exclusion Criteria:

* Medical diagnosis of asthma
* Significant condition or disease other than COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the standardized area under the curve for FEV1 (FEV1 AUC0-3) over the 3-hour assessment period at End Study (Week 6/ET). | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Hanania, MD, Principal Investigator — Baylor College of Medicine
Locations (19):
- United States (19):
  - Clinical Research Site, Mobile, Alabama
  - Clinical Research Site, Phoenix, Arizona
  - Clinical Research Site, DeLand, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Livonia, Michigan
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site, Albany, New York
  - Clinical Research Site, North Syracuse, New York
  - Clinical Research Site, Williamsville, New York
  - Clinical Research Site, Toledo, Ohio
  - Clinical Research Site, Medford, Oregon
  - Clinical Research Site, Portland, Oregon
  - Clinical Research Site, Greenville, South Carolina
  - Clinical Research Site, Spartanburg, South Carolina
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Abingdon, Virginia
  - Clinical Research Site, Richmond, Virginia
  - Clinical Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Result] Hanania NA, Boota A, Kerwin E, Tomlinson L, Denis-Mize K. Efficacy and safety of nebulized formoterol as add-on therapy in COPD patients receiving maintenance tiotropium bromide: Results from a 6-week, randomized, placebo-controlled, clinical trial. Drugs. 2009 Jun 18;69(9):1205-16. doi: 10.2165/00003495-200969090-00005. PMID 19537837